CLINICAL TRIAL: NCT04349761
Title: A Double-blind, Placebo-controlled, Randomized, First-in-human, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Oral Dose of MYMD1 Capsules in Healthy Male Adult Subjects
Brief Title: Single Ascending-dose Study to Evaluate Safety, Tolerability, and PK of MYMD1 in Healthy Male Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TNF Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MyMD-PK-001
Record Dates: First submitted 2020-02-10; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Undefined
Keywords: Pharmacokinetics; Phase I; First-in-Human; Safety; Tolerability; Hashimoto thyroiditis; Autoimmune
MeSH Terms: conditions — Hashimoto Disease

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, single ascending dose study.
Who Masked: Participant, Investigator
Masking Description: Placebo is identical in appearance to IP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 - 5mg MyMD1 (Experimental): 8 subjects randomized to receive either 5mg MyMD1 (6 subjects) or Placebo (2 subjects)
  Interventions: Drug: MyMD1; Drug: Placebo
- Cohort 2 - 10mg MyMD1 (Experimental): 8 subjects randomized to receive either 10mg MyMD1 (6 subjects) or Placebo (2 subjects)
  Interventions: Drug: MyMD1; Drug: Placebo
- Cohort 3 - 15mg MyMD1 (Experimental): 8 subjects randomized to receive either 15mg MyMD1 (6 subjects) or Placebo (2 subjects)
  Interventions: Drug: MyMD1; Drug: Placebo
- Cohort 4 - 20mg MyMD1 (Experimental): 8 subjects randomized to receive either 20mg MyMD1 (6 subjects) or Placebo (2 subjects)
  Interventions: Drug: MyMD1; Drug: Placebo
- Cohort 5 - 25mg MyMD1 or Placebo (Experimental): 8 subjects randomized to receive either 25mg MyMD1 (6 subjects) or Placebo (2 subjects)
  Interventions: Drug: MyMD1; Drug: Placebo

INTERVENTIONS:
Drug: MyMD1 — Isomyosamine 5mg capsules
Drug: Placebo — Placebo

SUMMARY:
Double-blind, placebo-controlled, First-in-Human, single ascending-dose study. Approximately 40 healthy adult male subjects will be given a single capsule of MYMD1 to determine its safety, how well it is tolerated, how the body acts on the experimental drug, and how the experimental drug acts on the body. This will be based on blood and urine sample analysis and other physical measurements.

DETAILED DESCRIPTION:
A single-center, double-blind, placebo-controlled, first-in-human, single ascending-dose study to evaluate the safety, tolerability, and pharmacokinetics of single oral dose capsules of MYMD1 in healthy male adult subjects. Each subject will participate in the study for approximately 7 weeks, including a Screening period of up to 30 days, a confinement period of 4 days, and a follow-up period of approximately 2 weeks. In each cohort, 8 subjects will be administered a single dose of either MYMD1 (N=6 in each cohort) or Placebo (N=2 in each cohort), under fasted conditions, and each subject will participate in only 1 of the 5 cohorts during the study. Anticipated dosing levels will be 5mg (Cohort 1), 10mg (Cohort 2), 15mg (Cohort 3), 20mg (Cohort 4), and 25mg (Cohort 5). Sentinel dosing will be used to initiate each cohort, and the first 2 subjects will be randomized 1:1 to receive either MYMD1 or Placebo. The remaining subjects will be dosed 5:1 to receive either MYMD1 or Placebo, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent.
* Stable medical history and general health.
* Body weight between 60 - 100 kg and Body Mass Index (BMI) of 18-31 kg/m2.
* Estimated GFR (eGFR) - mL/min/1.73m2 or estimated creatinine clearance (CLcr) (mL) ≥90.
* Normal hepatic function.
* Adequate peripheral venous access.
* Test negative for HIV, hepatitis C virus antibodies, and hepatitis B surface antigen (HBsAg).
* Test negative for drugs of abuse.
* Willing and able to complete all study assessments and procedures and to communicate effectively with the Investigator and study center staff.
* Willing to use effective contraception from Day -1 until 90 days after receiving study medication.

Exclusion Criteria:

* Allergy to any product ingredients.
* Unable to swallow capsules.
* Elective medical procedure during study.
* Abusing drugs or alcohol and/or history of drug or alcohol dependence within 6 months of study entry.
* History of seizure disorder requiring medical treatment after 18 years of age.
* Current smoker or smokeless tobacco user.
* Participation in drug or medical device clinical study within 30 days of study. entry or 5 times half-life of study drug, whichever is longer.
* Medically significant standard clinical laboratory assessments.
* Significant medical condition which might interfere with the study or put subject at significant risk.
* QTcF >450 ms or clinically significant ECG abnormalities.
* Elevation of blood pressure (BP) - Supine BP >145mmHg; Diastolic BP. >92mmHg;l heart rate (HR) >100 bpm.
* Gastrointestinal malabsorption.
* Abnormal thyroid function (TSH, T4 and/or T3 levels): elevated thyroid antibodies (anti- TPO and/or anti-Thyroglobulin); thyroid goiter, or known thyroid nodule(s) at Baseline; >Abnormal renal function (estimated GFR >90mL/min/1.73m2 or estimated creatinine clearance <90mL) and/or abnormal hepatic function at Baseline.
* Treatment with any prescription or nonprescription drugs, including vitamins, minerals, or herbal and dietary supplements, within 14 days or 5 half-lives of Day 1, whichever is longer - except Tylenol.
* Use within 30 days prior to Day 1 of any drugs or substances, including grapefruit juice, that are known to strongly inhibit or induce cytochrome P450 (CYP) enzymes.
* Donation of blood or blood product within 56 days of Day 1.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 5 days
  Any untoward medical occurrence in a subject which does not necessarily have a causal relationship with this treatment. Assessed as number and percent of patients with adverse events, compared across treatment and Placebo groups .
Changes in Physical examination: Neurologic Systems | 5 days
  Neurologic systems, including testing of patellar reflex using rubber mallet. Assessed by Investigator, based on education, experience, and training, as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Variation of MyMD1 concentration in blood plasma as a function of time | 5 days
  AUC (0-inf)
Change from Baseline QTcF and QTcB | 5 days
  Derived from centrally-overread 12-lead ECGs, measured in triplicate, based on Holter monitoring. Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Number of Patients with Changes in clinical laboratory values - Serum Chemistry: BUN, Creatinine, Glucose, Magnesium, Cholesterol, Calcium, Uric Acid, C-Reactive Protein, Total Bilirubin, Direct Bilirubin, Phosphate, and Triglycerides. | 5 days
  Number of patients with clinically significant changes from Baseline in Blood Urea Nitrogen (BUN); Creatinine; Glucose (fasting); Magnesium; Cholesterol; Calcium; Uric Acid; C-Reactive Protein; Total Bilirubin; Direct Bilirubin; Phosphate; and Triglycerides, compared across treatment and Placebo groups.
  All tests measured in mg/dL.
Percentage of Patients with Changes in clinical laboratory values - Serum Chemistry: BUN, Creatinine, Glucose, Magnesium, Cholesterol, Calcium, Uric Acid, C-Reactive Protein, Total Bilirubin, Direct Bilirubin, Phosphate, and Triglycerides. | 5 days
  Percentage of patients with clinically significant changes from Baseline in Blood Urea Nitrogen (BUN); Creatinine; Glucose (fasting); Magnesium; Cholesterol; Calcium; Uric Acid; C-Reactive Protein; Total Bilirubin; Direct Bilirubin; Phosphate; and Triglycerides, compared across treatment and Placebo groups.
  All tests measured in mg/dL.
Number of Patients with Changes in clinical laboratory values - Serum Chemistry: albumin, globulin, Total protein. | 5 days
  Number of patients with clinically significant changes from Baseline in albumin, globulin, and total protein, compared across treatment and Placebo groups. All tests measured in g/dL.
Percentage of Patients with Changes in clinical laboratory values - Serum Chemistry: albumin, globulin, Total protein. | 5 days
  Percentage of patients with clinically significant changes from Baseline in albumin, globulin, and total protein, compared across treatment and Placebo groups. All tests measured in g/dL.
Number of Patients with Changes in clinical laboratory values - Serum Chemistry: Electrolytes | 5 days
  Number of patients with clinically significant changes from Baseline in Potassium, Sodium, Chloride, and Carbon Dioxide (bicarbonate), compared across treatment and Placebo groups. All tests measured in mmol/L.
Percentage of Patients with Changes in clinical laboratory values - Serum Chemistry: Electrolytes | 5 days
  Percentage of patients with clinically significant changes from Baseline in Potassium, Sodium, Chloride, and Carbon Dioxide (bicarbonate), compared across treatment and Placebo groups. All tests measured in mmol/L.
Number of Patients with Changes in clinical laboratory values - Serum Chemistry: Creatine Kinase muscle/brain (MB) fraction | 5 days
  Number of patients with clinically significant changes from Baseline in Creatine Kinase muscle/brain (MB) fraction, compared across treatment and Placebo groups. All tests measured in ng/mL.
Percentage of Patients with Changes in clinical laboratory values - Serum Chemistry: Creatine Kinase muscle/brain (MB) fraction | 5 days
  Percentage of patients with clinically significant changes from Baseline in Creatine Kinase muscle/brain (MB) fraction, compared across treatment and Placebo groups. All tests measured in ng/mL.
Number of Patients with Changes in clinical laboratory values - Serum Chemistry: Gamma Glutamyl Transferase, Lactate dehydrogenase, Aspartate Aminotransferase, Alanine aminotransferase, Alkaline phosphatase, Creatine kinase, and Amylase | 5 days
  Number of patients with clinically significant changes from Baseline in Gamma Glutamyl Transferase, Lactate dehydrogenase, Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT), Alkaline phosphatase, Creatine kinase, and Amylase,compared across treatment and Placebo groups. All tests measured in U/L.
Percentage of Patients with Changes in clinical laboratory values - Serum Chemistry: Gamma Glutamyl Transferase, Lactate dehydrogenase, Aspartate Aminotransferase, Alanine aminotransferase, Alkaline phosphatase, Creatine kinase, and Amylase | 5 days
  Percentage of patients with clinically significant changes from Baseline in Gamma Glutamyl Transferase, Lactate dehydrogenase, Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT), Alkaline phosphatase, Creatine kinase, and Amylase,compared across treatment and Placebo groups. All tests measured in U/L.
Number of Patients with Changes in clinical laboratory values - Hematology:Red Blood Cell count | 5 days
  Number of patients with clinically significant changes from Baseline in Red Blood Cell count, compared across treatment and Placebo groups. All tests measured in Millions/microL.
Percentage of Patients with Changes in clinical laboratory values - Hematology:Red Blood Cell count | 5 days
  Percentage of patients with clinically significant changes from Baseline in Red Blood Cell count, compared across treatment and Placebo groups. All tests measured in Millions/microL.
Number of Patients with Changes in clinical laboratory values - Hematology: Platelet count, White Blood Cell count | 5 days
  Number of patients with clinically significant changes from Baseline in Platelet count and White Blood Cell count, compared across treatment and Placebo groups. All tests measured in Thousands/microL.
Percentage of Patients with Changes in clinical laboratory values - Hematology: Platelet count, White Blood Cell count | 5 days
  Percentage of patients with clinically significant changes from Baseline in Platelet count and White Blood Cell count, compared across treatment and Placebo groups. All tests measured in Thousands/microL.
Number of Patients with Changes in clinical laboratory values - Hematology: Hematocrit, Reticulocytes | 5 days
  Number of patients with clinically significant changes from Baseline in hematocrit and reticulocytes, compared across treatment and Placebo groups. All tests measured in %.
Percentage of Patients with Changes in clinical laboratory values - Hematology: Hematocrit, Reticulocytes | 5 days
  Percentage of patients with clinically significant changes from Baseline in hematocrit and reticulocytes, compared across treatment and Placebo groups. All tests measured in %.
Number of Patients with Changes in clinical laboratory values - Hematology: Mean corpuscular volume, Absolute Neutrophils, Absolute Lymphocytes, Absolute Monocytes, Absolute Eosinophils, and Absolute Basophils | 5 days
  Number of patients with clinically significant changes from Baseline in Absolute Neutrophils, Absolute Lymphocytes, Absolute Monocytes, Absolute Eosinophils, and Absolute Basophils, compared across treatment and Placebo groups. All tests measured in cells/microL.
Percentage of Patients with Changes in clinical laboratory values - Hematology: Mean corpuscular volume, Absolute Neutrophils, Absolute Lymphocytes, Absolute Monocytes, Absolute Eosinophils, and Absolute Basophils | 5 days
  Percentage of patients with clinically significant changes from Baseline in Absolute Neutrophils, Absolute Lymphocytes, Absolute Monocytes, Absolute Eosinophils, and Absolute Basophils, compared across treatment and Placebo groups. All tests measured in cells/microL.
Number of Patients with Changes in clinical laboratory values - Hematology: Mean corpuscular hemoglobin | 5 days
  Number of patients with clinically significant changes from Baseline in Mean corpuscular hemoglobin, compared across treatment and Placebo groups. All tests measured in pg.
Percentage of Patients with Changes in clinical laboratory values - Hematology: Mean corpuscular hemoglobin | 5 days
  Percentage of patients with clinically significant changes from Baseline in Mean corpuscular hemoglobin, compared across treatment and Placebo groups. All tests measured in pg.
Number of Patients with Changes in clinical laboratory values - coagulation: Fibrinogen | 5 days
  Number of patients with clinically significant changes from Baseline in fibrinogen (mg/dL), compared across treatment and Placebo groups.
Percentage of Patients with Changes in clinical laboratory values - coagulation: Fibrinogen | 5 days
  Percentage of patients with clinically significant changes from Baseline in fibrinogen (mg/dL), compared across treatment and Placebo groups.
Number of Patients with Changes in clinical laboratory values - coagulation: Prothrombin time, Activated partial thromboplastin time, Thrombin time | 5 days
  Number of patients with clinically significant changes from Baseline time, Activated partial thromboplastin time, Thrombin time compared across treatment and Placebo groups. All tests measured in seconds (sec).
Percentage of Patients with Changes in clinical laboratory values - coagulation: Prothrombin time, Activated partial thromboplastin time, Thrombin time | 5 days
  Percentage of patients with clinically significant changes from Baseline time, Activated partial thromboplastin time, Thrombin time compared across treatment and Placebo groups. All tests measured in seconds (sec).
Changes in Physical examination: Cardiovascular | 5 days
  Assessed by Investigator, based on education, training, and experience, using stethoscope, as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: Head, eye, ear, nose, and throat | 5 days
  Otolaryngologic head, eye, ear, nose, and throat exam, based on Investigator observation, based on experience, education, and training. Visual assessment of clinical appearance. Ear examined using a flashlight. Throat examined using a tongue depressor. Assessed by Investigator as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Electrocardiogram (ECG): Heart Rate | 5 days
  12-lead; Number of patients with clinically significant changes from Baseline in Electrocardiogram (ECG) measures of Heart Rate (beats per minute - bpm). Assessed by Investigator as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms"
Changes in Electrocardiogram (ECG): PR, RR, QRS, QT, QTcF, and QTcB | Time of Assessment (24-Hour Clock)
  12-lead. Number of patients with changes from Baseline in PR Interval (ms); RR Intermal (ms); QRS Interval (ms); QT Interval (ms); QTcF Interval (ms); and QTcB Interval (ms)
Vital signs: Oral Temperature (degrees Centigrade) | 5 days
  Oral temperature, using oral thermometer. Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: General Appearance | 5 days
  Physical signs and symptoms assessed by Investigator observation, based on experience, education, and training. May include observation of obesity or dermatologic conditions. Assessed by Investigator as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: Respiratory | 5 days
  Respiratory, measured in breaths per minute (bpm) Assessed by Investigator, based on education, experience, and training, as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: Gastrointestinal | 5 days
  Gastrointestinal signs and symptoms. May include evaluation of normal bowel movements or abdominal pain. Assessed by Investigator, based on education, experience, and training, as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: Body Weight | 5 days
  Body Weight measured in kg using scale. Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: Height | 5 days
  Height (cm) measured using ruler attached to weighing scale.
Pharmacokinetics: AUC | 5 days
  Area Under the Curve (AUC) (0-last): variation of a drug concentration in blood plasma as a function of time
Pharmacokinetics: Cmax | 5 days
  Cmax - Maximum Concentration of drug substance in blood plasma
Pharmacokinetics: tmax | 5 days
  tmax - Time to Maximum Concentration of drug substance in blood plasma
Pharmacokinetics: t 1/2 | 5 days
  Time to metabolism of 1/2 of dose (eg, half-life) of drug substance in blood plasma
Pharmacokinetics: CL/F | 5 days
  Oral Clearance of the drug substance (CL/F)
Pharmacokinetics: V2/F | 5 days
  V2/F
Vital Signs: Pulse Rate | 5 days
  pulse rate measured in beats per minute (bpm). Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Vital signs: Blood Pressure | 5 days
  Sitting diastolic and systolic blood pressure, measured by Karotkoff Cuff in mmHg. Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Vital signs: Respiratory Rate | 5 days
  Respiratory rate, measured in breaths per minute. Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Thyroid Test: Trilodothyronine (Free T3) | 5 days
  Number and percent of patients with clinically significant changes from Baseline in Free T3 (pg/mL), compared across treatment and Placebo groups.
Thyroid Test: Thyroxine (Free T4) | 5 days
  Number and percent of patients with clinically significant changes from Baseline in Free T4 (ng/dL), compared across treatment and Placebo groups.
Thyroid Test: Thyroid Stimulating Hormone (TSH) | 5 days
  Number and percent of patients with clinically significant changes from Baseline in TSH (mIU/L), compared across treatment and Placebo groups.
Urinalysis: Urobilinogen | 5 days
  Number and percent of patients with clinically significant changes from Baseline in Urobilinogen (eu/dL), compared across treatment and Placebo groups.
Urinalysis (Microscopic) | 5 days
  Number and percent of patients with clinically significant changes from Baseline in Red Blood Cell (RBC), Epithelial Cells, Bacteria, Casts, and White Blood Cell (WBC) counts, compared across treatment and Placebo groups. All units measured as /lpf.

OTHER OUTCOMES:
Biomarker assessment: TNF alpha | 5 days
  Tissue Necrosis Factor (TNF) alpha
Biomarker assessment: thyroglobulin | 5 days
  thyroglobulin (IU/mL)
Biomarker assessment: TPO antibodies | 5 days
  thyroperoxidase (TPO) antibodies
Biomarker assessment | 5 days
  pyridyloxobutyl (POB) adducts in hemophilia

CONTACTS AND LOCATIONS:
Overall Officials: Art Simon, PhD, Study Director — Palm Beach CRO, LLC; Leonard J Dunn, MD, Principal Investigator — Clinical Research of West Florida
Locations (1):
- Palm Beach CRO, LLC, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No